CLINICAL TRIAL: NCT01131000
Title: A Multicenter, Randomized, Double-blind, Parallel, Placebo-controlled Trial To Evaluate The Efficacy, Safety, and Pharmacokinetics of Ibuprofen Injection in Adult Febrile Patients
Brief Title: Efficacy, Safety, and Pharmacokinetics of Intravenous Ibuprofen in Adult Febrile Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: A. J. Kazimi, Chief Executive Office, Cumberland Pharmaceuticals Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPI-CL-004
Record Dates: First submitted 2010-05-24; First posted 2010-05-26 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2010-05

CONDITIONS: Fever
MeSH Terms: conditions — Fever | interventions — Ibuprofen; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ibuprofen (Experimental)
  Interventions: Drug: Ibuprofen
- Saline (Placebo Comparator): Normal Saline
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Ibuprofen — Intravenous ibuprofen, 100 mg, Single-dose
  Arms: Ibuprofen
Drug: Ibuprofen — Intravenous ibuprofen, 200mg, single dose
  Arms: Ibuprofen
Drug: Ibuprofen — Intravenous ibuprofen, 400 mg, Single-dose
  Arms: Ibuprofen
Other: Normal Saline — Normal Saline, 100 ml, Single-dose
  Other Names: 0.9 % NaCL; 0.9 % Sodium Chloride
  Arms: Saline

SUMMARY:
The primary objective of this study is to evaluate the efficacy of intravenous ibuprofen on reducing fever at 4 hours.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy of a single 400 mg dose of intravenous ibuprofen on reducing fever greater than or equal to 101.0ºF (38.3ºC), as compared with the efficacy of parallel placebo treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Be hospitalized
2. Have new (not chronic, within last 7 days) onset of fever, documented by temperature greater than or equal to 101.0ºF (38.3ºC)
3. Have adequate intravenous access
4. Have the ability to understand the requirements of the study, be willing to provide written informed consent (as evidenced by signature on an informed consent document approved by an Institutional Review Board), and agree to abide by the study restrictions and to return for the required assessments

Exclusion Criteria:

1. Be less than 18 years of age
2. Have received antipyretic drug therapy (e.g., aspirin, other NSAIDs, or acetaminophen) within 4 hours before dosing
3. Have any history of allergy or hypersensitivity to any component of IVIb, NSAIDs (including aspirin), or COX-2 inhibitors
4. Be pregnant or nursing
5. Have a history of severe head trauma that required current hospitalization, intracranial surgery, or stroke within the previous 30 days, or any history of intracerebral arteriovenous malformation, cerebral aneurysm, or central nervous system mass lesions
6. Weigh less than 40 kg
7. Have a history of congenital bleeding diatheses (e.g., hemophilia) or any active clinically significant bleeding, or have underlying platelet dysfunction, including (but not limited to) idiopathic thrombocytopenic purpura, disseminated intravascular coagulation, or congenital platelet dysfunction
8. Have gastrointestinal bleeding that has required medical intervention within the previous 6 weeks (unless definitive surgery has been performed)
9. Have a platelet count less than 30,000/mm3
10. Be receiving full dose anticoagulation therapy
11. Have fever secondary to blood or drug reaction
12. Have an expected life span of less than 14 days because of imminent withdrawal of life support or severity of illness
13. Be receiving treatment with corticosteroids (Patients who are expected to receive corticosteroids during the Treatment Period or through Hour 120 of the Post-treatment Period are not eligible.)
14. Have neurogenic fever
15. Be on dialysis, have oliguria or creatinine greater than 3.0 mg/dL, or be receiving nephrotoxic drugs
16. Have had major surgery within the past 12 hours, unless adequate hemostasis has been achieved
17. Have received another investigational drug within the past 30 days
18. Become afebrile (temperature below 101.0ºF [38.3ºC]) before dosing and not redevelop fever entry criteria during this hospitalization
19. Be otherwise unsuitable for the study, in the opinion of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2002-06; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Percent of patients with fever reduction to less than 101.0 degree fahrenheit following a single dose of intravenous ibuprofen. | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Bernard, M.D., Study Chair — Cumberland Pharmaceuticals, Inc.
Locations (11):
- United States (8):
  - Orlando Regional Medical Center, Orlando, Florida
  - Barnes Jewish Hospital, St Louis, Missouri
  - Moses H. Cone Memorial Hospital, Greensboro, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Methodist Healthcare - University Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Skyline Medical Center, Nashville, Tennessee
  - Ben Taub General Hospital, Houston, Texas
- Australia (2):
  - Newcastle Mater Misericordiae Hospital, New Lambton, New South Wales
  - Flinders Medical Centre, Adelaide, South Australia
- Mahidol University Siriraj Hospital, Bangkok, Thailand

REFERENCES:
- [Derived] Morris PE, Promes JT, Guntupalli KK, Wright PE, Arons MM. A multi-center, randomized, double-blind, parallel, placebo-controlled trial to evaluate the efficacy, safety, and pharmacokinetics of intravenous ibuprofen for the treatment of fever in critically ill and non-critically ill adults. Crit Care. 2010;14(3):R125. doi: 10.1186/cc9089. Epub 2010 Jun 30. PMID 20591173